CLINICAL TRIAL: NCT02215395
Title: Phase 1, Open-label Study to Evaluate the Effects of Concurrent Administration of Vaginal Antimycotic Medication (Miconazole Nitrate) on the Pharmacokinetics of Nestorone and Ethinyl Estradiol Delivered by a Contraceptive Vaginal Ring Releasing a Daily Dose of 150 ug of NES and 15 ug of EE
Brief Title: An Open-label Study to Evaluate the Effects of Concurrent Administration of Vaginal Antimycotic Medication Miconazole Nitrate on the Pharmacokinetics of Nestorone and Ethinyl Estradiol Delivered by a Contraceptive Vaginal Ring in Normal Ovulating Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Population Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 571
Record Dates: First submitted 2014-05-29; First posted 2014-08-13 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Antifungal Drug Adverse Reaction
Keywords: Nestorone; miconazole nitrate
MeSH Terms: interventions — ST 1435; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CVR treatment cycle (Experimental): Women who meet all inclusion and no exclusion criteria will be randomized to the first treatment cycle with the CVR alone followed by the second treatment cycle with the CVR and miconazole (one of three dosing regimens) or the first treatment cycle with the CVR and miconazole followed by the second treatment cycle with the CVR alone.
  Interventions: Drug: NES/EE CVR

INTERVENTIONS:
Drug: NES/EE CVR — Concurrent administration of vaginal antimycotic medication (Miconazole Nitrate) on the pharmacokinetics of Nestorone (NES) and ethinyl estradiol (EE) delivered by a contraceptive vaginal ring (CVR)
  Other Names: Nestorone (NES) and ethinyl estradiol (EE) delivered by a contraceptive vaginal ring (CVR)

SUMMARY:
To evaluate the pharmacokinetics (PK) of EE and NES released from the CVR in the presence of a single dose and multiple doses of antimycotic co-medication (miconazole nitrate suppository or cream).

ELIGIBILITY:
Inclusion Criteria:

* Healthy women, inclusive of ages 18-35* years at the enrollment visit
* Intact uterus and both ovaries
* Prior history of regular menstrual cycles that usually occur every 28 ± 7 days when not using hormonal contraception; if postpartum or post-abortal, history of regular menstrual cycles of 21-35 days in length and resumption of at least one cycle with a cycle length consistent with her past cycles
* In the opinion of the investigator, able to comply with the protocol, e.g. live within the study site catchment area or within a reasonable distance from the study site
* May be sterilized or at risk of becoming pregnant
* Willing to use a non-hormonal method of contraception for one month prior to the initial insertion of the NES/EE CVR and the one month washout period
* Willing to abstain from sexual intercourse during the miconazole nitrate treatment period(s)
* Signed informed consent prior to entry into the trial

Exclusion Criteria:

* Known hypersensitivity to estrogens or progestins
* Pregnant, trying to become pregnant, or breastfeeding
* Known hypersensitivity to silicone rubber
* Undiagnosed abnormal vaginal bleeding
* Undiagnosed vaginal discharge, vaginal lesions or abnormalities. Subjects diagnosed at screening with a Chlamydia or gonococcus infection may be included in the trial following treatment; partner treatment is also recommended. Investigators should make a determination if subjects are at high risk for reinfection, e.g., multiple sex partners, untreated partner, and whether such subjects can be included
* History of pelvic inflammatory disease since the subject's last pregnancy
* History of toxic shock syndrome
* In accordance with the Bethesda system of classification: Women with a current (within the last 20 months) abnormal Pap smear suggestive of high-grade pre-cancerous lesion (s), including HGSIL
* Cystoceles or rectoceles or other anatomical abnormality that would preclude use of a vaginal ring
* Women planning to undergo major surgery during the trial
* Women who smoke 15 cigarettes or more per day must be evaluated by the PI for inclusion based on risk factors that would increase their risk for cardiovascular disease and thromboembolism, e.g., lipid levels, glucose level, BP, BMI, family history of cardiovascular disease at a young age
* Current or past thrombophlebitis or thromboembolic disorders
* History of venous thrombosis or embolism in a first-degree relative, <55 years of age suggesting a familial defect in the blood coagulation system, which in the opinion of the PI, suggests that use of a hormonal contraceptive could pose a significant risk
* Cerebrovascular or cardiovascular disease
* History of retinal vascular lesions, unexplained partial or complete loss of vision
* Known or suspected carcinoma of the breast
* Carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasia
* Past history of any other carcinoma unless in remission for more than five years
* Current or history of medically diagnosed severe depression, which, in the opinion of the investigator, could be exacerbated by the use of a hormonal contraceptive
* Headaches with focal neurological symptoms
* Severe constipation in the opinion of the investigator
* History of cholestatic jaundice of pregnancy or jaundice with prior steroid use
* Benign or malignant liver tumors; active liver disease
* Diastolic blood pressure (BP) >85 mm Hg and/or systolic BP >135 mm Hg after 5-10 minutes rest (at screening)
* Known or suspected alcoholism or drug abuse within their lifetime
* Elevated serum fasting clinical chemistry values or complete blood count (CBC) values designated clinically significant by the investigator and/or medically qualified sub-investigator
* Screening hemoglobin levels less than 12.5 g/dL or hematocrit less than 38%.
* Participation in another clinical trial involving an investigational drug within the last 30 days (prior to screening)
* BMI >29
* Use of liver enzyme inducers on a regular basis
* Use of monthly injectable contraceptives, unless suspended 2 months before initiation of the treatment. Use of Depo-Provera [depo-medroxyprogesterone (DMPA)] unless suspended 6 months before treatment
* Current use of implanted hormonal contraceptives, including Mirena [progestin containing intrauterine system (IUS)], Jadelle, Norplant, Implanon or Nexplanon (if now available in the USA).**
* Known HIV, Hepatitis B or Hepatitis C infection
* History of frequent vaginal infections in the opinion of the investigator

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Drug Drug Interaction of NES/EE CVR and topical anti-fungal medication | Week 12
  To evaluate adverse reactions to a topical anti-fungal medication when used in conjunction with the NES/EE CVR

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Morrison, MD, Principal Investigator — QPS-Biokinetic
Locations (1):
- QPS Bio-Kinetic, Springfield, Missouri, United States

REFERENCES:
- [Derived] Simmons KB, Kumar N, Plagianos M, Roberts K, Hoskin E, Han L, Alami M, Creasy G, Variano B, Merkatz R. Effects of concurrent vaginal miconazole treatment on the absorption and exposure of Nestorone(R) (segesterone acetate) and ethinyl estradiol delivered from a contraceptive vaginal ring: a randomized, crossover drug-drug interaction study. Contraception. 2018 Mar;97(3):270-276. doi: 10.1016/j.contraception.2017.10.010. Epub 2017 Oct 31. PMID 29097225